CLINICAL TRIAL: NCT05938959
Title: Erector Spinae Plane Block for Pediatric Idiopathic Scoliosis Surgery. A Prospective, Randomized, Double-blinded Clinical Trial.
Brief Title: Erector Spinae Plane Block for Pediatric Idiopathic Scoliosis Surgery
Acronym: ESPB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3/2023
Record Dates: First submitted 2023-05-24; First posted 2023-07-11 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Scoliosis Idiopathic
Keywords: pain management; peripheral nerve block; erector spinae plane block; euromonitoring
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will be randomly allocated to receive ultrasound-guided ESP block with 0,2% ropivacaine or ESP block with the sham block by computer software 1:1. A researcher who will not be involved in the study will prepare the randomization list and concealed group assignments in consecutively numbered, sealed, opaque envelopes. A consultant anesthesiologist will follow management to open the envelopes shortly before the nerve block performance to reveal the group allocation and perform the procedure according to the assignment. The surgeon, patients, and anesthesia team will be masked to the study group. Group blinding unmasking will only occur once the statistical analysis is complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham group (Active Comparator): Bilateral ESPB under ultrasound guidance bi-level Th3-6 and Th9-L1(adjusted to the incision line): 0.3-0.5ml/kg 0,9% Normal Saline
  Interventions: Drug: Sham block
- ESPB group (Active Comparator): Bilateral ESPB under ultrasound guidance bi-level Th3-6 and Th9-L1(adjusted to the incision line): 0.3-0.5ml/kg 0.2% Ropivacaine (max 2.5mg/kg)
  Interventions: Drug: ESPB

INTERVENTIONS:
Drug: Sham block — Bilateral ESPB under ultrasound guidance bi-level Th3-6 and Th9-L1(adjusted to the incision line): 0.3-0.5ml/kg 0,9% normal saline
  Other Names: 0,9% normal saline
  Arms: Sham group
Drug: ESPB — Bilateral ESPB under ultrasound guidance bi-level Th3-6 and Th9-L1(adjusted to the incision line): 0.3-0.5ml/kg 0.2% Ropivacaine (max 2.5mg/kg)
  Other Names: 0,2% ropivacaine
  Arms: ESPB group

SUMMARY:
The study aims to assess the effect of the interfacial plane blocks on the pain level, the course of postoperative rehabilitation, and its anti-inflammatory analgesic effect.

DETAILED DESCRIPTION:
This study evaluates the analgesic efficacy in adolescents of bilevel, bilateral erector spinae plane (ESP) blocks after posterior spinal fusion surgery by assessing postoperative pain scores and opiate requirements as the primary outcome measures. We aim to investigate how ESP blocks, performed under ultrasound guidance at the two vertebral levels, contribute to postoperative pain control. This will be determined by measuring numerical rating pain scores repeatedly following surgery and opiate consumption until the patient is discharged from the hospital. These primary outcome measures will be compared between a treatment group of participants receiving ESP blocks and a control group receiving a sham block. Our primary hypothesis is that ESP blocks significantly reduce postoperative pain and opiate requirements.

ELIGIBILITY:
Inclusion Criteria:

* age 10-18 years old
* pediatric patients who will undergo the surgical correction of idiopathic scoliosis

Exclusion Criteria:

* a history of chronic pain (use of gabapentin/pregabalin for > 3 months or opioid use > 1 repeated opioid prescription in the last three months)
* morbid obesity (BMI > 99th percentile)
* previous surgery
* back abnormalities
* infection at block application area
* coagulopathy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain Numerical Rating Scale | 30 minutes after surgery
  Pain Numerical Rating Scale (0 - no pain, 10 - the worst pain)
Pain Numerical Rating Scale | 60 minutes after surgery
  Pain Numerical Rating Scale (0 - no pain, 10 - the worst pain)
Pain Numerical Rating Scale | 90 minutes after surgery
  Pain Numerical Rating Scale (0 - no pain, 10 - the worst pain)
Pain Numerical Rating Scale | 120 minutes after surgery
  Pain Numerical Rating Scale (0 - no pain, 10 - the worst pain)
Pain Numerical Rating Scale | 6 hours after surgery
  Pain Numerical Rating Scale (0 - no pain, 10 - the worst pain)
Pain Numerical Rating Scale | 12 hours hours after surgery
  Pain Numerical Rating Scale (0 - no pain, 10 - the worst pain)
Pain Numerical Rating Scale | 24 hours after surgery
  Pain Numerical Rating Scale (0 - no pain, 10 - the worst pain)
Pain Numerical Rating Scale | 48 hours after surgery
  Pain Numerical Rating Scale (0 - no pain, 10 - the worst pain)

SECONDARY OUTCOMES:
neutrophil/lymphocyte ratio | 12 hours and 24 hours after surgery
  neutrophil/lymphocyte ratio
platelet/lymphocyte ratio | 12 hours and 24 hours after surgery
  platelet/lymphocyte ratio
Nausea or Vomiting | during first 24 hours after surgery
  presence or absence
total opioid consumption | Day 1 after surgery
  intravenous milligrams of morphine equivalents
total opioid consumption | Day 2 after surgery
  intravenous milligrams of morphine equivalents
total opioid consumption | Day 3 after surgery
  intravenous milligrams of morphine equivalents
total opioid consumption | Day 4 after surgery
  intravenous milligrams of morphine equivalents
total opioid consumption | Day 5 after surgery
  intravenous milligrams of morphine equivalents
total opioid consumption | Day 6 after surgery
  intravenous milligrams of morphine equivalents
total opioid consumption | Day 7 after surgery
  intravenous milligrams of morphine equivalents
Motor Evoked Potential amplitude | up to seven days prior to the correction of scoliosis
  Motor Evoked Potentials durring surgery
Motor Evoked Potential amplitude | up to 24 weeks following the correction of scoliosis
  Motor Evoked Potentials during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Kotwicki, Ph.D., Study Director — Poznań University of Medical Sciences
Locations (2):
- Poland (2):
  - Department of Spine Diseases and Pediatric Orthopedics, University of Medical Sciences, Poznań, Poland, Poznan, Wielkopolska
  - Poznan University of Medical Sciences, Poznan